CLINICAL TRIAL: NCT03344302
Title: Oxytocin Administration During Cesarean Section Before Versus After Fetal Delivery Randomized Clinical Trial
Brief Title: Oxytocin Administration During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OACS
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 100 women were assigned to receive an intravenous infusion of oxytocin 30 units in a rate 125 mL/hour minutes diluted into 500 mL of normal 0.9% sodium chloride) immediately after opening the visceral peritoneum just before incising the uterine wall during Cesarean section
  Interventions: Drug: Oxytocin
- Control group (Active Comparator): 100 women were assigned to an intravenous infusion of oxytocin 30 units in a rate 125 mL/hour diluted into 500 mL of normal 0.9% sodium chloride) immediately after clamping the umbilical cord during cesarean section
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — intravenous infusion of oxytocin 30 units over 5 minutes diluted into 500 mL of normal 0.9% sodium chloride

SUMMARY:
Cesarean delivery is defined as fetal birth through incisions in the abdominal wall and the uterine wall. This definition does not include removal of the fetus from the abdominal cavity in the case of uterine rupture or in the case of an abdominal pregnancy The guidelines of the Royal College of Obstetricians and Gynaecologists on caesarean section recommend a slow intravenous bolus dose of 5 IU of oxytocin after delivery of the infant. Intravenous oxytocin has a short half life (4-10 minutes); therefore the potential advantage of an oxytocin infusion at caesarean section is in maintaining uterine contractility throughout the surgical procedure and immediate postpartum period, when most primary haemorrhage occurs

ELIGIBILITY:
Inclusion Criteria:

* Primigravida or multigravida
* Term (37 - 42 weeks),
* Singleton pregnancies
* Booked for elective caesarean section.
* Accepting to participate in the study.

Exclusion Criteria:

* • Medical disorders involving the heart, liver, kidney or brain.

  * Diabetes mellitus and hypertension.
  * Blood disorders (e.g. coagulopathies, thrombocytopenia)
  * Patients requiring blood transfusion due to anemia.
  * Risk factors for uterine atony e.g. macrosomia, polyhydramnios and multiple pregnancy.
  * Previous 2 or more cesarean section
  * Placenta previa or placental abruption
  * Previous major obstetric haemorrhage (>1000 ml) in previous deliveries.
  * Known fibroid or adenomyosis.
  * Women who received anticoagulant therapy.
  * Severe preeclampsis.
  * Uterine anomalies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
rate of blood loss | 4 hours
  collection of the blood in the drape below the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided